CLINICAL TRIAL: NCT05864144
Title: A Phase 1/2, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SNS-101 (Anti VISTA) as Monotherapy and in Combination With Cemiplimab in Patients With Advanced Solid Tumors
Brief Title: A Study of SNS-101 (Anti VISTA) Monotherapy and in Combination With Cemiplimab in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sensei Biotherapeutics, Inc. (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNS-101-2-1
Record Dates: First submitted 2023-04-21; First posted 2023-05-18 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor, Adult; Advanced Solid Tumor; Head and Neck Cancer; Breast Cancer; Colon Cancer; Pancreatic Cancer; Gastric Cancer; Esophageal Cancer; Prostate Cancer; Uterine Cancer; Cervix Cancer; Ovarian Cancer; Kidney Cancer; Bladder Cancer; Thyroid Cancer; Melanoma; Sarcoma; Advanced Cancer; Metastatic Cancer; Refractory Cancer; Non Small Cell Lung Cancer; Merkel Cell Carcinoma
Keywords: Solnerstotug
MeSH Terms: conditions — Head and Neck Neoplasms; Breast Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Prostatic Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms; Thyroid Neoplasms; Melanoma; Sarcoma; Neoplasm Metastasis; Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Merkel Cell | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - SNS-101 Monotherapy Dose Escalation and Dose Expansion (Experimental): SNS-101 IV alone every 21 days. Patients will initially enroll in dose escalation cohorts.
  Interventions: Drug: SNS-101 (anti-VISTA)
- Part B - SNS-101 in combination with cemiplimab and Dose Expansion (Experimental): SNS-101 IV and cemiplimab IV every 21 days. Patients will initially enroll in dose escalation cohorts.
  Interventions: Drug: SNS-101 (anti-VISTA); Drug: Cemiplimab
- Part C - Cohort Expansion - SNS-101 alone or in combination with cemiplimab (Experimental): SNS-101 IV alone or in combination with cemplimab IV every 21 days at the RP2D.
  Interventions: Drug: SNS-101 (anti-VISTA); Drug: Cemiplimab

INTERVENTIONS:
Drug: SNS-101 (anti-VISTA) — SNS-101 IV every 21 days.
Drug: Cemiplimab — Cemiplimab IV every 21 days.
  Arms: Part B - SNS-101 in combination with cemiplimab and Dose Expansion; Part C - Cohort Expansion - SNS-101 alone or in combination with cemiplimab

SUMMARY:
Phase 1/2 study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of SNS-101, a novel anti VISTA IgG1 monoclonal antibody as monotherapy or in combination with cemiplimab in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1/2 open-label, multi-center, dose escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of SNS-101, a novel anti VISTA IgG1 monoclonal antibody as monotherapy or in combination with cemiplimab in patients with advanced solid tumors.

This study is being conducted in three parts:

* Part A: Phase 1 Monotherapy Dose Escalation and Dose Expansion (SNS-101 alone)
* Part B: Phase 1 Combination Dose Escalation and Dose Expansion (SNS-101 in combination with cemiplimab)
* Part C: Phase 2 Cohort Expansion (SNS-101 alone or in combination with cemiplimab)

Once the dose escalation portion is complete enrollment will expand to targeted tumor types:

* Approximately 10 patients with colorectal cancer (CRC) will be enrolled in the Monotherapy Dose Expansion.

  o Additional tumor types and doses may be considered upon consultation with the Sponsor.
* Approximately 50 patients with CRC, head and neck cancer (H&N), melanoma, and non-small cell lung cancer (NSCLC) will be enrolled in the Combination Dose Expansion.

  * A minimum of 8 and a maximum of 10 CRC patients will be enrolled in the Combination Dose Expansion.
  * Additional tumor types and doses may be considered upon consultation with the Sponsor.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically documented locally advanced, unresectable or metastatic solid tumor.
* Having received and failed or was intolerant to standard of care for advanced disease or not eligible for standard of care therapy with the following tumor types for patients in Phase 1 dose expansion cohorts:

  1. Microsatellite Stable (MSS) CRC (both monotherapy and combination cohorts); no more than 3 lines of prior systemic therapy for metastatic disease.
  2. H&N cancer (combination cohort only); no more than 2 lines of prior systemic therapy for metastatic disease.
  3. Melanoma (combination cohort only); no more than 3 lines of prior systemic therapy for metastatic disease, including at least 1 prior treatment with a BRAF inhibitor for patients with a BRAF mutation.
  4. NSCLC (combination cohort only); no more than 2 lines of prior systemic therapy for metastatic disease, including at least 1 prior treatment with a targeted therapy for patients with a mutation such as EGFR, ALK, KRAS, or RET.
  5. Patients with H&N cancer, melanoma, and NSCLC (or additional tumor types that typically respond to PD1/PD-L1 monotherapy) must have received a prior PD1/PD-L1 where best response was stable disease and progression occurred during treatment or within 3 months of last dose of PD1/PD-L1.

Additional tumor types and doses may be considered.

* Measurable disease
* ECOG performance status 0 or 1.
* Life expectancy of ≥ 3 months.
* Willing to provide pre-treatment (archival or fresh) and on-treatment tumor biopsy samples.
* Adequate organ function
* Women of childbearing potential and fertile males with WOCBP partners must use highly effective contraception during the study and for 180 days after the study. Patients must agree not to donate eggs (ova, oocytes) or sperm during the study.

Key Exclusion Criteria:

* Use of anti-PD-1/PD-L1 targeting monoclonal antibody therapy, monoclonal antibody therapy, chemotherapy, biologic, investigational, or radiotherapy within 2 weeks of Cycle 1 Day 1.
* Clinically significant unresolved toxicities from prior anticancer therapy.
* Grade 3 or higher immune-related adverse event on prior PD-1/PD-L1 blockade or prior agents targeting stimulatory or co-inhibitory T cell receptor.
* Known other previous/current malignancy requiring treatment within ≤ 2 years except for limited disease treated with curative intent, such as carcinoma in situ, squamous or basal cell skin carcinoma, or superficial bladder carcinoma.
* Known asymptomatic or symptomatic brain metastasis or leptomeningeal disease.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events - Part A & B | Day 1 through 90 days after the last dose
  Incidence, nature and severity of treatment-related adverse events
Determine the Recommended Phase 2 dose or maximum tolerated dose - Part A & B | Approximately 15 months
  Incidence and nature of dose-limiting toxicities
Objective Response Rate (ORR) - Part C | Day 1 through study completion (approximately 1 year)
  Measured by RECIST 1.1 and iRECIST

SECONDARY OUTCOMES:
Determine pharmacokinetic profile (maximum concentration) of SNS-101 - Part A, B & C | Day 1 through 30 days after the last dose
  Measured by maximum concentration
Determine pharmacokinetic profile (area under the curve) of SNS-101 - Part A, B & C | Day 1 through 30 days after the last dose
  Measured by area under the curve
Determine pharmacokinetic profile (total clearance) of SNS-101 - Part A, B & C | Day 1 through 30 days after the last dose
  Measured by total clearance
Determine pharmacokinetic profile (terminal half life) of SNS-101 - Part A, B & C | Day 1 through 30 days after the last dose
  Measured by serum terminal half-life
Number of participants with anti-SNS-101 antibodies post-administration of SNS-101 - Part A, B & C | Day 1 through 30 days after the last dose
  Measured by anti-SNS-101 neutralizing anti-drug antibodies
Objective Response Rate (ORR) - Part A & B | Day 1 through study completion (approximately 1 year)
  Measured by RECIST 1.1 and iRECIST
Duration of Response (DoR) - Part A, B & C | Day 1 through study completion (approximately 1 year)
  Measured by RECIST 1.1 and iRECIST
Disease Control Rate (DCR) - Part A, B & C | Day 1 through study completion (approximately 1 year)
  Measured by RECIST 1.1 and iRECIST
Progression Free Survival - Part A, B and C | Day 1 through study completion - approximately 1 year (Part A, B & C)
  Measured by RECIST 1.1 and iRECIST
Adverse Events - Part C | Day 1 through study completion (approximately 1 year)
  Incidence, nature and severity of treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ron Weitzman, MD, Study Director — Sensei Biotherapeutics, Inc.
Locations (10):
- United States (10):
  - UCLA Hematology/Oncology, Los Angeles, California
  - University of Colorado Cancer Center - Anschutz Medical, Aurora, Colorado
  - Norton Healthcare, Louisville, Kentucky
  - Henry Ford Cancer, Detroit, Michigan
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - University of Pennsylvania, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - NEXT Oncology Dallas, Irving, Texas
  - South Texas Accelerated Research Therapeutics (START) San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No